CLINICAL TRIAL: NCT01666925
Title: Efficacy Study of ChAd63MVA ME-TRAP Prime-boost Vaccination Against Plasmodium Falciparum Infection.
Brief Title: Efficacy of Malaria Vaccines in Kenyan Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC046
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ChAd63 ME-TRAP and MVA ME-TRAP (Experimental): ChAd63 ME-TRAP / MVA ME-TRAP heterologous prime-boost immunisation
  Interventions: Biological: ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation
- Rabies vaccine (Active Comparator): 2 x 2.5IU Verorab
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation — ChAd63 ME-TRAP: 5 x 10^10vp MVA ME-TRAP: 2 x 10^8 pfu
  Arms: ChAd63 ME-TRAP and MVA ME-TRAP
Biological: Rabies vaccine — 2 x 2.5IU Verorab
  Other Names: Verorab
  Arms: Rabies vaccine

SUMMARY:
Malaria transmission is falling in some parts of Africa as bed nets and anti-malarials become more widely available. However, transmission still persists and it appears that additional control measures are required. The leading malaria vaccine candidate in development is RTS,S which has efficacy against clinical malaria measured at 30-50% in the field. This partial protection might be enhanced by combination with other components. The other vaccination approach that has produced repeatable efficacy in humans is the use of viral vectors to induce T cell responses. Previous attempts with this vaccine approach have been effective in challenge studies in Oxford, but ineffective in the field, probably because of reduced immunogenicity.

Recently, studies in Oxford, Kenya and the Gambia have shown higher levels of immunogenicity by using a chimpanzee adenovirus (ChAd63) followed by an attenuated vaccinia virus (modified vaccinia Ankara) to deliver the pre-erythrocytic antigen, multiple epitope string with thrombospondin- related adhesion protein (ME-TRAP).

The increase in immunogenicity has lead to sterile protection in 3 out of 14 volunteers and partial protection in 5 out of 14 volunteers in challenge studies.

The investigators propose a Phase 2b study of 120 healthy adult men in Kenya. The investigators will assess the efficacy and further evaluate the immunogenicity and safety profile of the vaccine regimen. The investigators also intend to assess the correlates of efficacy and natural immunity.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult males aged 18 - 50 years in good health.
* Will remain resident in the study area for the study duration.
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Informed Consent

Exclusion Criteria:

* Any significant medical disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Hypersensitivity to Verorab, the trial vaccines or the antimalarial used.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, kathon, neomycin
* History of splenectomy.
* Haemoglobin less than 10.0 g/dl
* Clinically significant abnormalities of laboratory screening tests (full blood count, ALT, creatinine levels).
* Blood transfusion within the month preceding enrolment.
* History of vaccination with previous experimental malaria vaccines or other vaccines likely to impact on findings of study (e.g. other MVA or adenovirus vectored vaccines)
* Administration of any other vaccine or immunoglobulin within 2 weeks before vaccination.
* HIV or Hepatitis B surface antigen seropositivity.
* Current participation in another clinical trial or recent participation within 12 weeks of this study.
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Vaccine Efficacy | 18 weeks
  The first episode of P.falciparum infection positive by PCR, for P.falciparum.

SECONDARY OUTCOMES:
Vaccine immunogenicity | 24 weeks
  Measures of immunogenicity will include:
  Ex vivo ELISPOT responses to overlapping pools of ME - TRAP peptides. Cultured ELISPOT responses to overlapping pools of ME - TRAP peptides. ICS by flow cytometry for cell mediated immune responses ELISA for antibodies to malaria antigens
Reactogenicity | 24 weeks
  All solicited and unsolicited local and systemic vaccine- linked adverse events (AEs) including clinically significant laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI/Wellcome Trust Programme, Centre for Geographic Medicine Research - Coast, Kilifi, Kenya